CLINICAL TRIAL: NCT00621972
Title: A Prospective Observational Study on the Use of Iodinated Contrast for AV Fistula Salvage in Stage 4/5 CKD Using Bicarbonate Prophylaxis
Brief Title: AV Fistula Salvage in Advanced CKD Using Sodium Bicarbonate Prophylaxis
Status: Withdrawn | Type: Observational
Sponsor: MaineHealth (Other)
Responsible Party: Sponsor
Other Study IDs: MMC3230; 0200.178070
Record Dates: First submitted 2008-02-12; First posted 2008-02-22 (Estimated); Last update posted 2018-09-20 (Actual); Status verified 2018-09

CONDITIONS: Acute Renal Failure
Keywords: acute renal failure; arteriovenous fistula; KIM-1; chronic kidney disease
MeSH Terms: conditions — Acute Kidney Injury; Arteriovenous Fistula; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observation: Chronic kidney disease patients presenting for fisulta evaluation with documented GFR<30ml/min by abbreviated MDRD calculation.

SUMMARY:
This is an observational study assessing the impact of conventional dose iodinated contrast on the renal function of advanced chronic kidney disease patients undergoing arteriovenous fistula evaluation using a standard sodium bicarbonate prophylaxis protocol. In addition, this model allows for pre and post procedure measurements of kidney function, providing a unique opportunity to assess the utility of novel biomarkers for contrast-induced kidney injury.

Our primary hypothesis is that there will be no change in serum creatinine post-procedure when using a standard sodium bicarbonate prophylaxis protocol. Our secondary hypothesis is that there will be no change in urinary kidney-injury marker-1 (KIM-1) post-procedure using a standard sodium bicarbonate prophylaxis protocol. In addition, we will assess the impact of different patient characteristics on the development of contrast-induced kidney injury, such as diabetes, coronary artery disease, hypertension, and angiotensin converting enzyme inhibitor therapy.

DETAILED DESCRIPTION:
The National Kidney Foundation publishes kidney disease outcome guidelines for improving care of the chronic kidney disease (CKD) patient. Regarding hemodialysis vascular access, the recommendation is for early placement of an arteriovenous fistula (AVF) to improve morbidity and mortality outcomes, specifically when the glomerular filtration rate is less than 25ml/min, corresponding to stage 4 and 5 CKD. Despite its advantages, the need for surveillance of the AVF to determine maturation for use and maintain optimal longevity requires the use of interventional procedures. While radiocontrast use can lead to acute, often reversible kidney injury, its use in AVF evaluation has renewed interest with the recent implication of gadolinium-enhanced MRI being associated with a rare disorder of skin swelling and induration called nephrogenic systemic fibrosis. CKD patients are particularly susceptible to long term adverse outcomes from contrast-induced kidney injury, with 1 year mortality in stage 4 and 5 CKD patients being 44% and 62%, respectively. While optimal fluid therapy to prevent contrast-induced kidney injury remains uncertain, several prospective randomized trials using sodium bicarbonate pretreatment have shown a lower incidence of contrast-related kidney injury compared to isotonic saline. Traditional markers of acute kidney injury, including serum creatinine, blood urea nitrogen, and creatinine clearance have been insensitive in differentiating contrast-induced kidney injury from other forms of renal injury. Kidney injury marker-1 (KIM-1) is a transmembrane receptor induced to very high levels in the proximal tubule of the nephron following ischemic and nephrotoxic injury. KIM-1 has been shown in a small cohort of patients to differentiate ischemic kidney injury from other forms of acute and chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* >18 yrs age
* chronic kidney disease, documented GFR<30ml/min by abbreviated MDRD calculation

Exclusion Criteria:

* Inpatients
* Pediatric patients
* Non-English speaking patients
* established dialysis patients
* patients receiving iodinated contrast within 30 days of current procedure
* patients with central arterial manipulation within 30 days of current procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stage 4 and 5 chronic kidney disease patients with AV fistula placed but have not initiated dialysis.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-01; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Assess the impact of conventional dose iodinated contrast on the renal function of stage 4 and 5 chronic kidney disease patients undergoing arteriovenous fistula evaluation using a standard sodium bicarbonate prophylaxis protocol. | 48 hours

SECONDARY OUTCOMES:
Assess the impact of conventional dose iodinated contrast on urinary kidney injury marker-1 (KIM-1) levels. | 3 hours and 48 hours
Assess the impact of different patient characteristics on the development of contrast-induced kidney injury, such as diabetes, coronary artery disease, hypertension, and angiotensin converting enzyme inhibitor therapy. | Baseline patient charcteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Scott M Benson, D.O., Principal Investigator — Maine Medical Center - Division of Nephrology
Locations (1):
- Maine Medical Center - Brighton Campus, Portland, Maine, United States